CLINICAL TRIAL: NCT04210375
Title: A Randomized, Double-Blind, Placebo-controlled, Single-ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of JK07 in Subjects With Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: Study of JK07 in Subjects With Heart Failure With Reduced Ejection Fraction (HFrEF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Salubris Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JK07.1.01
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; HFrEF; neuregulin 1; NRG-1; heregulin; HER3; HER4; ErbB3; ErbB4; reduced ejection fraction
MeSH Terms: conditions — Heart Failure; Fibromatosis, Gingival, 2

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, single-ascending dose with single active sentinel subject per cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JK07 (Active Comparator): Single dose of JK07 administered by intravenous infusion over 60 minutes
  Interventions: Drug: JK07
- Matching Placebo (Placebo Comparator): Single dose of placebo administered by intravenous infusion over 60 minutes
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: JK07 — Recombinant fusion protein consisting of a fully humanized immunoglobulin G1 monoclonal antibody and an active polypeptide fragment of the human growth factor NRG-1
  Arms: JK07
Drug: Matching Placebo — Vehicle control
  Arms: Matching Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-ascending dose study to assess the safety, tolerability, immunogenicity, PK, and exploratory efficacy of JK07 in subjects 18 to 80 years of age with HFrEF ≤40%.

Initially 5 cohorts are planned with the option to expand the study to a total of 7 cohorts. The size of the cohorts will range from 5 to 9 subjects. Each cohort will include one single active unblinded sentinel subject receiving a single IV dose of JK07 prior to randomized single dose administration of JK07 or placebo [3:1] in the remainder of the cohort.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-ascending dose study to assess the safety, tolerability, immunogenicity, PK, and exploratory efficacy of JK07 in HF subjects 18 to 80 years of age with LVEF ≤40%. Subjects must have been maintained on an optimal HF medical regimen for at least 2 months prior to enrollment and remain on the same treatment regimen throughout the course of the study, per the 2017 ACC/AHA/HFSA) treatment guidelines.

At screening, eligible subjects will undergo a physical examination, 2-dimensional transthoracic echocardiography (2D-TTE), ECG assessment, blood sampling for laboratory parameters, and urine testing. Safety assessments at screening will include hematology, biochemistry, coagulation, liver, and thyroid function.

Subjects will be observed in the hospital on continuous telemetry from the time of hospital admission until shortly before discharge approximately 48 hours later. During this time, they will additionally have safety labs, vital signs, PK and biomarker samples collected, and ECGs and 2D-TTEs performed.

Only a single dose of the investigational product will be administered and only a single hospital admission is planned per subject during the study. Subjects will complete follow-up visits through 180 days after administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 and 80 years with stable NYHA Class II or III HF diagnosis (ischemic or non-ischemic confirmed by medical history) at least 6 months prior to enrollment as confirmed by medical history.
2. Stable HF defined as no hospitalizations for cardiac-related issues within the previous 2 months prior to the screening visit or between screening and randomization, other than for routine percutaneous procedures such as device, battery, generator changes or pacemaker lead insertion/ replacement.
3. Subjects with clearly interpretable echocardiographic images and with a screening LVEF ≤ 40% in the absence of ≥ Grade 3 valvular disease on 2D-TTE.
4. Subjects must be taking clinician-directed appropriate pharmacological therapy for HF as per the 2017 ACC/AHA/HFSA treatment guidelines at stable doses and at investigator determined discretion (except for diuretics) for at least 2 months prior to informed consent.
5. Subjects with implantable cardioverter-defibrillators (ICDs) are allowed at the discretion of the investigator, but only if both the following criteria are met: (a) paced beats cannot exceed 15% of beats as quantified by screening e-Patch, and (b) if a non-paced baseline ECG can be obtained on day 1 prior to study drug administration.

5. Body mass index ≥18 kg/m2 and ≤45 kg/m2. 6. Screening hemoglobin ≥9.0 g/dL, platelets ≥100 K/mL, ANC ≥1500/mL. 7. Able and willing to use adequate contraception until the end of the study.

8. Capable of providing informed consent and to comply with the protocol.

Exclusion Criteria:

1. Participating in any other study, have received any other investigational drug within 30 days prior to screening or 5-half-lives or any other investigational implanted device within 30 days prior to screening, or are taking part in a nonmedication study which, in the opinion of the Investigator, would interfere with study compliance or outcome assessments.
2. Any past participation in a study that has investigated the NRG-1 pathway (e.g., Neucardin, Cimaglermin).
3. Heart failure due to hypertrophic cardiomyopathy, restrictive cardiomyopathy, arrhythmogenic right ventricula dysplasia (ARVD), stress-induced ("Takotsubo") cardiomyopathy, chemotherapy-induced cardiomyopathy, peripartum cardiomyopathy, infiltrative or inflammatory cardiomyopathies, and primary valvular disease.
4. Medically documented acute coronary syndrome within 3 months of screening or a medically documented acute MI within 6 months of screening.
5. Cardiac surgery, coronary artery revascularization, percutaneous coronary intervention, or valvuloplasty within 3 months prior to screening.
6. Any subject who has received an indication for coronary revascularization within 3 months prior to screening.
7. Any major surgical procedure within 1 month prior to screening or planned surgical procedure during the study period.
8. Sustained systolic blood pressure <90 mm Hg and/or diastolic blood pressure <50 mm Hg.
9. Sustained resting heart rate >100 beats per minute sustained for >15 minutes except in sustained atrial fibrillation when a heart rate of up to 110 beats per minute is acceptable.
10. Cerebrovascular accident or hospitalizations for CV (cardiovascular) causes other than routine percutaneous procedures such as device, battery, generator changes or pacemaker lead insertion/ replacement or device generator changes, including HF, chest pain, stroke, transient ischemic attack, or arrhythmias within 3 months prior to randomization.
11. At screening have an abnormal or clinically significant 12-lead ECG abnormality that, in the opinion of the Investigator, would affect efficacy or safety evaluation or place the subject at risk.
12. History or evidence of clinically significant arrhythmia uncontrolled by drug therapy or use of an implantable defibrillator, long QT syndrome, or evidence of QT prolongation with QTcF >450 ms for males or QTcF >470 ms for females prior to randomization.
13. Clinically significant renal dysfunction as measured by the estimated GFR <45 mL/min/1.73m2 at screening, or a clinically significant change in renal function between screening and baseline.
14. Clinically significant liver dysfunction as measured by: ALT >2.0 × ULN, alkaline phosphatase > 2.0 × ULN, AST >2.0 × the ULN, or GGT >2.0 × the ULN or serum bilirubin ≥ 1.2 × the ULN at screening, or a clinically significant change in liver function between screening and baseline.
15. Subjects with alteration of the coagulation panel (INR) and/or PT ≥ 1.5 × the ULN; aPTT ≥ 1.5 × ULN, or serum albumin ≤ 3 gm/dL. For subjects on warfarin or other anticoagulants, an INR (or PT) considered by the Principal Investigator as therapeutically appropriate will be allowed.
16. Subjects with values of CPK and/or CK-MB >2.5 times normal institutional limits at screening.
17. Any subject who by Investigator's judgement, has a significant hematuria or proteinuria at screening.
18. Concurrent treatment with Class Ia or III antiarrhythmic drugs (the medication must have been discontinued more than 2 months before informed consent).
19. Positive screening for HIV antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies.
20. Known history of or active alcohol abuse (no more than 14 units/week for males or 7 units/week for females) or use of illicit drugs within 1 year prior to randomization (excluding recreational use of marijuana or cannabidiol [CBD]-based products.
21. Other medical or psychiatric condition that, in the opinion of the Investigator, would preclude obtaining voluntary consent/assent or would confound the secondary objectives of study.
22. A history of pathologically-confirmed malignancy of any type or any pathologically-confirmed pre-malignant condition (e.g. ductal carcinoma in situ, colonic polyp with premalignant diagnosis, or cervical atypia).
23. Pregnant or lactating female subjects at screening.
24. Subjects with clinically significant or poorly controlled disease including, but not limited to, endocrine (including diabetes and thyroid) disease, neurological or psychiatric (even mild), GI, hematological, urological, immunological, or ophthalmic diseases as determined by the Investigator.
25. Subjects who are not non-smokers or light smokers (no more than 5 cigarettes per day) and who cannot abstain from smoking from 2 weeks prior to the administration of IP through the end of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Stanford University Medical Center, Stanford, California
  - Harvard Medical School/ Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Science University Hospital, Portland, Oregon
  - University of Texas Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang WHW, Steiner J, Kassi M, Wheeler MT, Spahillari A, Sweitzer NK, Grodin JL, Solomon N, Singhal S, McEwen AMG, Murphy SL. Single Ascending-Dose Study of Selective ErbB4 Agonist JK07 in Heart Failure With Reduced Ejection Fraction. JACC Basic Transl Sci. 2025 Sep;10(9):101352. doi: 10.1016/j.jacbts.2025.101352. Epub 2025 Jul 29. PMID 40737710

RESULTS

PARTICIPANT FLOW:
Groups:
- JK07 - Cohort 1: Experimental: JK07 0.03 mg/kg
  Cohort 1: Participants were administered 0.03 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
  JK07: Recombinant fusion protein consisting of a fully humanized immunoglobulin G1 monoclonal antibody and an active polypeptide fragment of the human growth factor NRG-1
- JK07 - Cohort 2: Experimental: JK07 0.09 mg/kg
  Cohort 2: Participants were administered 0.09 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
  JK07: Recombinant fusion protein consisting of a fully humanized immunoglobulin G1 monoclonal antibody and an active polypeptide fragment of the human growth factor NRG-1
- JK07 - Cohort 3: Experimental: JK07 0.27 mg/kg
  Cohort 3: Participants were administered 0.27 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
  JK07: Recombinant fusion protein consisting of a fully humanized immunoglobulin G1 monoclonal antibody and an active polypeptide fragment of the human growth factor NRG-1
- Matching Placebo: Matching Placebo: Vehicle control
  Single dose of placebo administered by intravenous infusion over 60 minutes, with 180 days of follow-up.
Period: Overall Study
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3 | Matching Placebo
Started | 4 | 4 | 3 | 3
Completed | 4 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was an ascending dose phase 1 trial. Participants were enrolled in an ascending fashion lower to higher doses of JK07.
Groups:
- JK07 - Cohort 1: Experimental: JK07 0.03 mg/kg
  Cohort 1: Participants were administered 0.03 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
- JK07 - Cohort 2: Experimental: JK07 0.09 mg/kg
  Cohort 2: Participants were administered 0.09 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
- JK07 - Cohort 3: Experimental: JK07 0.27 mg/kg
  Cohort 3: Participants were administered 0.27 mg/kg of JK07 single dose by intravenous infusion over 60 minutes, with 180 days of follow-up.
- Total: Total of all reporting groups
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3 | Matching Placebo | Total
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 1 | 3 | 10
  >=65 years | 0 | 2 | 2 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.9) | 61.3 (9.74) | 61.0 (14.93) | 54.3 (5.13) | 57.4 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 4
  Male | 4 | 2 | 2 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 4 | 3 | 3 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-emergent Adverse Events [Safety and Tolerability]
Description: All safety information is collected and evaluated.
Time Frame: Screening to 30 days
Population: All randomized participants
Measure: Number; unit: number of events
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3 | Matching Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 3
number of events
  Treatment emergent AEs | 4 | 3 | 8 | 2
  SAEs | 0 | 0 | 1 | 0

2. Secondary Outcome: AUC(0-last) of JK07
Description: Area under the concentration (time curve to the last quantifiable concentration) from blood samples taken on Days 1-4, and Days 7, 11, 15, 22, 30, and 60.
Time Frame: Baseline to 60 days
Population: All randomized participants were included in the noncompartmental analysis of pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3
Number analyzed (Participants) | 4 | 4 | 3
h*ng/mL | 5310 (80.6) | 34400 (2.9) | 139000 (15.1)

3. Other Pre Specified Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: 2D-transthoracic echocardiography-derived LVEF
Time Frame: Screening to 180 days
Population: All randomized participants.
Measure: Mean (Full Range); unit: % of LVEF
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3 | Matching Placebo
Number analyzed (Participants) | 4 | 4 | 3 | 3
% of LVEF
  Day 1 - pre dose | 34 [29 to 36] | 28 [21 to 32] | 25 [17 to 37] | 31 [28 to 37]
  Day 1 - 6 hrs post dose | 37 [34 to 39] | 30.5 [19 to 40] | 31 [23 to 35] | 33.7 [29 to 43]
  Day 2 | 39.8 [37 to 44] | 28.8 [21 to 41] | 30.7 [20 to 39] | 32.3 [32 to 33]
  Day 7 | 38.5 [29 to 51] | 33.5 [26 to 40] | 28 [21 to 37] | 27.3 [23 to 31]
  Day 15 | 42.5 [34 to 53] | 34.5 [28 to 40] | 28.3 [22 to 35] | 31 [27 to 38]
  Day 30 | 40.8 [33 to 49] | 33 [25 to 38] | 28.7 [20 to 38] | 32.7 [29 to 39]
  Day 60 | 38.5 [34 to 46] | 35.3 [28 to 44] | 30 [21 to 39] | 29.3 [22 to 33]
  Day 90 | 37 [30 to 51] | 36 [21 to 47] | 27 [16 to 39] | 25 [21 to 28]
  Day 135 | 36 [22 to 46] | 31.7 [26 to 39] | 32 [27 to 37] | 22 [19 to 25]
  Day 180 | 36 [33 to 40] | 38.7 [30 to 52] | 32.3 [24 to 44] | 33.7 [31 to 36]

4. Secondary Outcome: Cmax of JK07
Description: Maximum concentration from blood samples taken on Days 1-4, and Days 7, 11, 15, 22, 30, and 60.
Time Frame: Baseline to 60 days
Population: All randomized participants were included in the noncompartmental analysis of pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3
Number analyzed (Participants) | 4 | 4 | 3
ng/mL | 497 (44.3) | 1680 (20.9) | 5170 (13.8)

5. Secondary Outcome: t1/2 of JK07
Description: Half-life from blood samples taken on Days 1-4, and Days 7, 11, 15, 22, 30, and 60.
Time Frame: Baseline to 60 days
Population: All randomized participants were included in the noncompartmental analysis of pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3
Number analyzed (Participants) | 4 | 4 | 3
h | 8.11 (42.7) | 10.95 (10.8) | 18.32 (8.2)

ADVERSE EVENTS:
Time Frame: Entire study duration (~180 days)
Description: Subjects were observed for injection site reactions until Day 4 following IP administration, for DLAEs until Day 15 following IP administration, and for AEs and SAEs from the time of informed consent until 30 days after the IP administration. Following Day 30, only SAEs deemed at least possibly related to the study drug or study procedures were collected until the EOS visit (Day 180).
  AEs were graded using CTCAE v5.0.
Arm/Group | JK07 - Cohort 1 | JK07 - Cohort 2 | JK07 - Cohort 3 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 3/4 | 3/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JK07 - Cohort 1 (N=4) | JK07 - Cohort 2 (N=4) | JK07 - Cohort 3 (N=3) | Matching Placebo (N=3)
Upper Extremity Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — A single Grade 3 SAE of "upper extremity weakness" was reported in cohort 3. Subsequent to the upper extremity weakness, the subject experienced Grade 3 TEAE of brachial neuritis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JK07 - Cohort 1 (N=4) | JK07 - Cohort 2 (N=4) | JK07 - Cohort 3 (N=3) | Matching Placebo (N=3)
Mild heahache (Nervous system disorders) | 1 | 0 | 0 | 0
Moderate Headache (Nervous system disorders) | 1 (2) | 0 | 0 | 0
Change in vision (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Intermittent nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Muscle tightness in hips and left shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilateral shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Brachial neuritis of both upper extremities (Nervous system disorders) | 0 | 0 | 1 | 0
Elevated creatinine (Investigations) | 0 | 0 | 1 | 0
Myalgia and arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neuropathy exacerbation (Nervous system disorders) | 0 | 0 | 1 | 0
Elevated liver enzymes (Investigations) | 0 | 0 | 0 | 1
Left arm nerve pain (Nervous system disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This was a Phase 1, single ascending dose study intended to support the continued exploration of JK07 as a HF treatment. As such, these results provide only a very early picture of the potential safety profile and pharmacodynamics of JK07.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT04210375/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT04210375/SAP_001.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT04210375/ICF_002.pdf